CLINICAL TRIAL: NCT04735328
Title: Implementing Evidence-based PTSD Treatment in Adult Mental Health Clinics
Brief Title: Implementering PTSD Treatment
Acronym: ITV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian Center for Violence and Traumatic Stress Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ITV project Norway
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Post-traumatic Stress Disorder; Leadership; Implementation
Keywords: Implementation; Implementation strategy; Leadership; Organizational climate; Fidelity; PTSD treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: Participating clinics will be grouped in four groups - two groups will start the intervention in 2021, two groups will start in 2022. All participants receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): When clinics join the intervention, leaders will receive leadership training through the Leadership and Organizational Change for Implementation (LOCI) intervention.
  Therapists will receive training in evidence-based practices for treatment of Post-Traumatic Stress Symptoms (EMDR and CT-PTSD).
  Interventions: Behavioral: LOCI; Behavioral: CT-PTSD; Behavioral: EMDR

INTERVENTIONS:
Behavioral: LOCI — LOCI includes training of leaders in general leadership, implementation leadership, and implementation climate.
Behavioral: CT-PTSD — CT-PTSD (Cognitive Therapy for PTSD), treatment method developed for treating patients with Post Traumatic Stress Symptoms (PTSD).
Behavioral: EMDR — EMDR (Eye Movement and Desensitization Reprocessing), treatment method developed for treating patients with Post-Traumatic Stress Symptoms (PTSD).

SUMMARY:
The project will develop knowledge on how managers can lead the implementation of practices that have proven to be effective for post-traumatic stress disorders (PTSD) in adult specialized mental health services. Specifically, the project will examine the intervention named the Leadership and Organizational Change for Implementation (LOCI). This is an empirically and theoretically based innovation for implementation leadership that aims to support leaders in their organizational work of leading the implementation of EBPs in their clinics. It is hypothesized that the implementation of LOCI will improve leaders' general leadership qualifications, their implementation leadership qualifications, and the implementation climate in the clinics. Further, the investigators hypothesize that training in trauma screening will increase the amount of trauma screenings, moderated by the LOCI implementation, and also that training in trauma treatment will increase the amount of patients to be offered this kind of treatment, also moderated by the LOCI implementation.

DETAILED DESCRIPTION:
Leadership for implementation require leadership that supports effective implementation strategies at the organizational level. The Leadership and Organizational Change for Implementation (LOCI) is a leadership training program focusing on enhancing general leadership and implementation leadership in particular (Aarons, Ehrhart, Moullin, Torres, & Green, 2017). The aim of the project is to evaluate the implementation strategy used to implement evidence-based treatment for PTSD in adult specialized mental health services in Norway.

The Leadership and Organizational Change for Implementation (LOCI) consists of several components:

1. 360° assessment A 360° assessment where the LOCI leaders, the therapists who report to them, and the executive leader are asked to complete a web-based survey focused primarily on the leadership of the LOCI leader and the implementation climate in his/her unit. Questions to therapists and the executive leaders are worded so that they are reporting on the appropriate LOCI leader. The LOCI leaders are asked questions about their own leadership, climate in their clinic, and on the implementation citizenship of their therapists. Descriptive results from the 360° assessment are presented in an individual feedback report for each of the LOCI leaders in the LOCI condition. Each of the LOCI leaders will receive their own feedback reports during the initial and follow-up leadership trainings, and they will not be required to share it with anyone besides the research group. Feedback reports for the executives will utilize data aggregated across all clinics within the respective health trusts. Executives will be presented with their feedback reports at initial and follow-up organizational strategy meetings (see below).

Leadership training 2.1 Training 2.1.1 Initial leadership training: The LOCI intervention begins with a two-day workshop for the LOCI leaders. The workshop addresses leadership in general, with a particular focus on the full-range leadership model, transactional leadership, and implementation leadership. The LOCI leaders are challenged to share own experiences and views on leadership, and examples of leadership styles are shared and discussed. Implementation climate is also addressed, with a focus on strategies leaders can use to support implementation of EBPs. Mid-way in the workshop at both day 1 and 2, the feedback reports from the 360° assessment will be shared individually with each of the LOCI leaders. The LOCI facilitator and the LOCI leader review the report together, identifying strengths and areas they would like to further develop. In a collaborative method, the LOCI facilitator and the LOCI leader draft that leader's individual leadership development plan wherein goals and committed actions are detailed to facilitate enhancement in their leadership and the implementation climate of their clinic.

2.1.2 Booster leadership training: The leadership training is followed by a one day booster session after 4 and 8 months. Before each booster session, a new 360° assessment will be completed, resulting in updated feedback reports, where the data is presented in graphs so that it is easy to see the development from the baseline assessment to the assessment at 4 and 8 months. The feedback report makes the basis for the leaders´ subsequent work with the individual leadership development plan. Organizational strategies, goals, and leadership are addressed through group discussions.

2.1.3 Graduation: At month 12, there will be a ritual to mark the completion of the program. Accomplishments are celebrated, challenges are addressed, and plans for further sustainment are shared.

2.2 Coaching calls with first-level leaders The LOCI leaders will participate in weekly brief consultation calls over the phone (10-30 minutes) with their LOCI facilitator where the goals are to give the leaders the opportunities to strategize methods for overcoming barriers to EBP implementation; to follow up on the leadership development plan; and to update the leadership development plan according to the work being done and new information. Once a month the individual calls are replaced with one-hour group consultation calls with all the LOCI leaders within the cohort.

2.3 Organizational strategy meetings (OSMs) LOCI leaders and executives meet with the LOCI facilitator(s) for 2 hours following the first leadership training. At this meeting, the LOCI leaders and executives will receive feedback from the 360° survey followed by the iterative development of an implementation climate development plan in light of the results from the survey. The subsequent meetings take place on a web conferencing platform at months 4, 8, and 12.

The executive will participate in brief (15-30 minutes) monthly telephone coaching calls with the LOCI facilitator where the focus is to follow up on the implementation climate development plan in light of the results from the 360° survey.

Evidence-based practices for post-traumatic stress disorders (PTSD) During the project, therapists will be trained in screening for and diagnosing PTSD, using evidence-based assessment tools. In addition, two well-documented EBPs for PTSD will be implemented in Norwegian specialized mental health services: 1) Eye Movement Desensitization and Reprocessing (EMDR) is an integrative eight-phased approach which is guided by the Adaptive Information Processing model (Shapiro & Laliotis, 2015). 2) Cognitive Therapy for PTSD (CT-PTSD) is based on a model assuming that PTSD develops if the traumatic event is processed in a way that maintains the experience of serious current threat (Ehlers & Clark, 2000).

Personnel in all clinics will receive training (2-3 hours) in screening for trauma and post-traumatic stress symptoms. A sample of therapists will receive three days of training in one of the specific practices (EMDR or CT-PTSD). The therapists will receive 10 hours of group consultation divided by 2 hours once a month for 5 months.

Methods:

A prospective design will be used. All participating clinics will receive the same LOCI intervention. The clinics will be allocated into groups of 6-7 clinics. Two groups will receive LOCI from April 2020 till June 2021. Two groups will receive LOCI from April 2021 till June 2022.

The project will consist of three groups of participants:

1. First-level leaders will participate in the LOCI innovation and complete 360 degrees surveys. In addition, executive leaders will participate in organizational structural meetings to support first-level leaders, in addition to completing the surveys.
2. All therapists in the participating clinics will participate in the training of PTSD screening and the surveys. A sample of therapists will be trained and supervised in PTSD treatment.
3. Patients that are referred to the clinics as normal, report traumatic experiences and fulfill the criteria for PTSD will be offered to participate in the study. They will receive PTSD treatment, and complete surveys in connection with the treatment sessions. The project aims at recruiting 12 mental health clinics in 2021 and 12 clinics in 2022 in specialized services from all over Norway. The clinics will be recruited via the four regional health trust, which will receive an invitation by e-mail.

Inclusion and exclusion criteria Adult outpatient clinics in specialized health services are included. All leaders and therapists in the clinics will be asked to participate in the surveys. Administrative personnel are excluded as most of the measures will not be applicable to these staff. Staff must be employees of the participating clinics. Leaders that do not agree to participate in the leadership training (LOCI) will not be eligible to participate. Patients (18-100 years) with PTSD will be asked to participate in the study by their therapist. There are no specific exclusion criteria, as the referrals should follow standard procedures within the clinics.

Fidelity Therapists will videotape (EMDR) or audiotape (CT-PTSD) all sessions in all cases. Randomly chosen therapy sessions for each therapist will be checked for fidelity. Students will be trained to assess five fidelity sessions per therapist.

The therapists will receive written fidelity feedbacks as soon as possible after the session has been video or audiotaped.

Data collection and management Data are collected from therapists, LOCI leaders, and executives at baseline, and at 4, 8, 12, and 16 months. The surveys are distributed by e-mail. Participants are not given any compensation for their participation. The therapist and LOCI leader survey takes on average 15-20 minutes to complete, whereas the executive survey takes on average 10 minutes to complete. Results from some of the scales will be shared with the LOCI leaders (MLQ, ILS, IC, EBPAS) and the executive leaders (IC, and EBPAS)) as part of the LOCI. Patients will fill out a questionnaire by iPad in connection with all therapy sessions. It takes on average 30 minutes to complete. Patients can receive trauma treatment even if they do not want to participate in the research. All data will be stored on the University center for sensitive data. Results from some of the scales will be shared with the therapist by a report function on the iPad.

Discussion Implementation of EBP can be challenging. Leaders in the health care system have the responsibility that the services provide effective treatments to a certain number of patients within a given time period. In order to increase the probability that patients will receive the most effective care for their symptoms, the leaders have to obtain effective strategies to promote the adoption of the evidence-based treatment. The LOCI intervention addresses leadership in general, implementation leadership in particular, and organizational strategies in order to support the implementation of EBP and sustainment over time. Available data suggest that LOCI is effective in supporting implementation of EBP through strengthening leadership and a positive implementation climate (Aarons et al., 2017). This study will examine the adaption of LOCI in a Norwegian mental health setting. We will examine whether the LOCI will have an effect on leadership, the implementation climate at the clinics, and the clinic´s ability to offer trauma-focused treatments to patients with elaborated levels of post-traumatic stress symptoms. The knowledge derived from this study can be used to support the implementation of other EBPs within the mental health system.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary child and adult specialized mental health clinics that agree to the terms and conditions of the project, that is training, recruitment of patients, and data collection.
* Patients with PTSD symptoms and that agree to participate in the project.

Exclusion Criteria:

* Clinics or patients that do not agree to the terms and the conditions of the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Implementation leadership scale (ILS) | 4 weeks
  ILS assesses the degree to which leaders are knowledgeable, proactive, perseverant, and supportive during evidencebased practice (EBP) implementation.Scored from 0 (not at all) to 4 (to a very great extent).

SECONDARY OUTCOMES:
Number of trauma assessments and patients that receive trauma treatment | 12 months
  Practitioners are asked to report the number of trauma assessments done within the last 4 months. The practitioners that have been trained in either TF-CBT, EMDR or CT-PTSD will also be asked to report the number of patients that receive the specific treatment.
The Multifactor Leadership Questionnaire (MLQ) | 12 months
  A 36-item measure addressing transformational and transactional leadership. Scored from 0 (not at all) to 4 (frequently, if not always)
The Implementation Climate (IC) | 12 months
  A 6-item measure addressing the implementation climate in the organization. Scored from 0 (not at all) to 4 (often, if not always).
Workload (QPS) | 12 months
  Thirteen items from the QPS Nordic questionnaire. Coping with work (6 items), job demands (7 items). Scored from 1 (very seldom or never) to 5 (very often or always).
The Implementation Citizenship Behavior Scale (ICBS) | 12 months
  A six-item measure addressing employee behaviour that goes beyond their duty to support the implementation of EBP.
  Scored from 0 (Not at all) to 4 (Frequently, if not always).
The Treatment integrity checklist for EMDR (T-TIP EMDR) | 12 months
  consists of 16 items evaluating whether the therapist carries out the manual correctly ("yes" or "not relevant" = 1 point, "no" = 0 point). Maximal score is 16 points.
Cognitive Therapy for Post-Traumatic Stress Disorder: A Checklist of Therapist Competency | 12 months
  consists of 16 items evaluating therapists' general and specific therapeutic skills on a range between 0 (poor) and 6 (excellent)
Stressful Life Events Screening Questionnaire - revised (SLESQ) | 12 months
  15 questions on stressful life events (0 = no, 1 = yes)
PTSD Checklist (PCL-5) | 12 months
  20 symptom items. A total symptom severity scale score ranging from 0 to 80. (0 = not at all, 4 = a lot)

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian Center for Violence and Traumatic Stress Studies (NKVTS), Oslo, Norway